CLINICAL TRIAL: NCT05355311
Title: L-carnitine Supplementation for Co-occurring Depression and Alcohol Use Disorder in Youth: An Open Trial Pilot Study
Brief Title: Enhancing the Effects of Alcohol Treatment With L-Carnitine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); Colorado State University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2101002877; R21AA029033-01A1 (NIH)
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: This study is an open-label study designed to assess the effects of L-carnitine supplementation on responses to in vivo alcohol cue exposure in the human laboratory setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-Carnitine (Experimental): L-carnitine is a nutritional supplement and emerging research shows it has neuroprotective properties and may help treat alcohol use disorder and depression, 2.97 g daily for 6 weeks
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — L-carnitine is an endogenous precursor of acetylcholine and metabolic intermediate that facilitates the transport of acetyl groups across the mitochondrial membrane and shows promise for treating alcohol use disorder and depression.

SUMMARY:
The primary objective of this study is to evaluate the effects of L-carnitine, 2.97g daily on alcohol cue-elicited alcohol craving during a human laboratory paradigm after 4 weeks of daily dosing among participants ages 18-25 with alcohol use disorder (AUD) as confirmed by the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5™) and who report at least mild depressive symptoms on the Beck Depression Inventory-II. Secondary objectives include evaluation of L-carnitine (2.97g/day) on alcohol craving and use, subjective effects of alcohol consumption, mood, sleep, alcohol use negative consequences, study retention, and safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 25 years old, inclusive
2. Self-report consuming alcohol ≥ 2 days/week on average in the past 28 days
3. Meets the DSM-5 criteria for alcohol use disorder (AUD)
4. Be interested in reducing alcohol use
5. Report at least mild depressive symptoms, as indicated by a score ≥ 14 on the Beck Depression Inventory II.
6. Be able to verbalize an understanding of the consent/assent form, able to provide written informed consent/assent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
7. Have parent permission, if younger than 18 years
8. Be able to take oral medication and be willing to adhere to the medication regimen
9. Complete all assessments required at screening and baseline.
10. Provide contact information of someone, such as a parent or other family member, who may be able to contact the subject in case of a missed appointment or follow-up assessment.
11. Agree to the schedule of visits, verbally acknowledge ability to attend each scheduled visit, participate in phone visits and report no scheduled events or a job that may substantially interfere with study participation.
12. Not anticipate any significant problems with transportation arrangements or available time to travel to the study site over the next 2 months.
13. Agree (if the subject's sex is female and of childbearing potential) to use at least one reliable method of birth control, unless subject is surgically sterile, partner is surgically sterile, or subject is postmenopausal. Examples of reliable methods include (but may not be limited to):

    1. oral contraceptives
    2. contraceptive sponge
    3. contraceptive skin patch
    4. double barrier diaphragm (diaphragm/spermicidal or condom/spermicidal)
    5. intrauterine contraceptive system
    6. levonorgestrel implant
    7. medroxyprogesterone acetate contraceptive injection
    8. complete abstinence from sexual intercourse
    9. hormonal vaginal contraceptive ring

Exclusion Criteria:

1. Be currently receiving alcohol use disorder treatment
2. Have significant alcohol withdrawal symptoms (score > 10) on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-AR)
3. Have a coexisting moderate to severe substance use disorder other than cannabis and nicotine, as defined by DSM-5 criteria
4. Have a urine toxicology screen positive performed during screening or baseline for any of the following substances:

   1. benzodiazepines
   2. cocaine
   3. opiates
   4. amphetamines
   5. buprenorphine
   6. methadone
   7. barbiturates
   8. oxycodone
   9. 3, 4-methylenedioxy-methamphetamine (MDMA, also known as ecstasy)
   10. methamphetamines
5. Have been treated with a pharmacotherapy for alcohol use disorder or a carbonic anhydrase inhibitor within 30 days prior to randomization
6. Compelled to alcohol treatment by the juvenile justice system or has probation or parole requirements that might interfere with study participation
7. Have a history of liver disease or have clinically significant abnormal laboratory values, including elevation of liver enzymes (AST, ALT) 5-fold above the upper limit of normal (ULN), or bilirubin greater than 2 times the upper limit of normal.
8. History of renal impairment or renal stones, heart problems or defects, abnormal blood pressure, progressive neurodegenerative disorder, or clinically significant neurological disorders
9. Clinically significant physical abnormalities per physical exam, hematological assessment, bilirubin concentration, or urinalysis
10. Pregnancy, nursing, or refusal to use reliable birth control, if female of childbearing potential
11. Stable dose of any prescribed psychotropic medication (i.e., no dose changes in the 2 months prior to randomization)
12. Current or lifetime diagnosis of psychotic disorders or current bipolar disorder
13. Current suicidality risk
14. Known sensitivity to acetyl-l-carnitine
15. Be a subject who in the opinion of the investigator could not be safely withdrawn from alcohol without medical detoxification
16. Have a serious or unstable medical illness or any potentially life-threatening or progressive medical condition other than addiction that may compromise subject safety or study conduct
17. Have abnormal calculated creatinine clearance defined as < 80 mL/min
18. Have data suggesting cirrhosis of the liver (albumin < 3.2 g/dL, or ascites by physical exam)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Alcohol Craving (derived from the Alcohol Urge Questionnaire; 0 to 20; higher scores = greater urge to drink) | Week 5
  Strength of self-reported alcohol craving

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miranda, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
With participant consent, data will be uploaded into appropriate NIH repository as required.
Time Frame: Within 12 months of publication
Access Criteria: Any investigator who requests access in writing will be provided with the requested information.